CLINICAL TRIAL: NCT06189716
Title: Evaluation of Gas Composition in the Oropharynx During High-flow Oxygen Therapy Through Nasal Cannula in Healthy Volunteers: a Physiological Study
Brief Title: Gas Composition in the Oropharynx During High-flow Oxygen Therapy Through Nasal Cannula in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: HFNC-OXIMETRY
Record Dates: First submitted 2023-12-19; First posted 2024-01-03 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2023-12

CONDITIONS: Healthy Volunteers
Keywords: healthy volunteers; HFNC; high flow oxygen; oximetry; capnometry; pharyngeal

STUDY DESIGN:
Intervention Model Description: Measurement of the inspiratory (FiO2) and expiratory (FeO2) fractions of oxygen (FiСO2 and FeСO2, respectively), as well as the inspiratory and expiratory fractions of carbon dioxide (FiСO2 and FeСO2, respectively) in the hypopharynx of healthy volunteers during high-flow oxygen therapy through nasal cannulas in different physiological conditions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental): High flow oxygen through nasal cannula, oxygen and carbon dioxide measurement in the hypopharynx
  Interventions: Device: High flow oxygen through nasal cannula

INTERVENTIONS:
Device: High flow oxygen through nasal cannula — High flow oxygen through nasal cannula and measurement of oxygen and carbon dioxide fraction in the hypopharynx of healthy volunteers in different physiological conditions.

SUMMARY:
Observational, randomized studies and their meta-analyses have shown the high effectiveness of high-flow oxygen therapy through nasal cannulas, reaching 50-60% in acute hypoxemic respiratory failure. Some bench studies showed the advantages of high-flow oxygen therapy compared with standard oxygen therapy, consisting in reducing the anatomical dead space and maintaining a given inspiratory oxygen fraction in the hypopharynx of the mannequin, but the actual state of the gas composition of the hypopharynx was not studied. The study aim is measurement of the inspiratory (FiO2) and expiratory (FeO2) fractions of oxygen, as well as the inspiratory (FiСO2) and expiratory (FeСO2) fractions of carbon dioxide in the hypopharynx of healthy volunteers during high-flow oxygen therapy through nasal cannulas in different physiological conditions.

DETAILED DESCRIPTION:
Randomized controlled trials showed reduction of tracheal intubation in high-flow oxygen therapy through nasal cannulas group in patients with acute respiratory failure as compared to standard oxygen therapy and noninvasive ventilation before Coronavirus disease-19 (COVID-19) pandemic.

The World Health Organization (WHO) declared the outbreak a pandemic of COVID-19 on March 11th, 2020. Since then observational, randomized studies and their meta-analyses have shown the high effectiveness of high-flow oxygen therapy through nasal cannulas (HFNC), reaching 50-60% in acute hypoxemic respiratory failure.

Bench studies showed the advantages of HFNC compared with standard oxygen therapy, consisting in reducing the anatomical dead space and maintaining a given inspiratory oxygen fraction in the hypopharynx of the mannequin, but the actual state of the gas composition of the hypopharynx during HFNC was not studied.

The study aim is measurement of the inspiratory (FiO2) and expiratory (FeO2) fractions of oxygen, as well as the inspiratory (FiСO2) and expiratory (FeСO2) fractions of carbon dioxide in the hypopharynx of healthy volunteers during high-flow oxygen therapy through nasal cannulas in different physiological conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers
* Age over 18 years
* Written informed consent.

Exclusion Criteria:

* Any primary or secondary lung diseases (COPD, bronchial asthma, interstitial lung diseases, metastatic lung disease, lung cancer)
* Any chronic diseases that can cause respiratory disorders (chronic heart failure, liver cirrhosis, systemic connective tissue diseases, cancer, neuromuscular diseases etc)
* Heart rhythm disturbances
* Body mass index more than 30 kg/m2
* Swallowing disorders
* History of epileptic syndrome
* Recent head surgery or anatomy that precludes the use of nasal cannulas
* Pregnancy and lactation period
* Inability to cooperate with staff.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-01-09 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Inspiratory oxygen fraction (FiO2) in the hypopharynx | 5 minutes
  Inspiratory oxygen fraction (FiO2) in the hypopharynx during different physiological conditions
Expiratory oxygen fraction (FeO2) in the hypopharynx | 5 minutes
  Expiratory oxygen fraction (FeO2) in the hypopharynx during different physiological conditions
Inspiratory fraction of carbon dioxide (FiCO2) in the hypopharynx | 5 minutes
  Inspiratory fraction of carbon dioxide (FiCO2) in the hypopharynx during different physiological conditions
Expiratory fraction of carbon dioxide (FeCO2) in the hypopharynx | 5 minutes
  Expiratory fraction of carbon dioxide (FeCO2) in the hypopharynx during different physiological conditions

SECONDARY OUTCOMES:
Respiratory rate (RR) | 5 minutes
  Respiratory rate (RR) during different physiological conditions
Tidal volume (VT) | 5 minutes
  Tidal volume (VT) during different physiological conditions
Peripheral oxygen saturation (SpO2) | 5 minutes
  Peripheral oxygen saturation (SpO2) during different physiological conditions
Modified ventilatory ratio (mVR) | 5 minutes
  Modified ventilatory ratio (mVR) during different physiological conditions. mVR = [RR * tidal volume* (PetCO2 (mmHg) - 4 mmHg)] / [predicted body weight (kg) * 100 * 37,5 mmHg]
The ratio of oxygen saturation by pulse oximetry/inspiratory oxygen fraction to respiratory rate (ROX-index) | 5 minutes
  ROX-index (SpO2/FiO2/RR) during different physiological conditions
Comfort | 5 minutes
  Visual-analog scale (VAS) for comfort evaluation (from 1 to 10, 1-full comfort, 10-full comfort)

CONTACTS AND LOCATIONS:
Overall Officials: Andrey I Yaroshetskiy, MD, PhD, ScD, Principal Investigator — I.M. Sechenov First Moscow State Medical University
Locations (1):
- Sechenov University Clinic#4, Moscow, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frat JP, Thille AW, Mercat A, Girault C, Ragot S, Perbet S, Prat G, Boulain T, Morawiec E, Cottereau A, Devaquet J, Nseir S, Razazi K, Mira JP, Argaud L, Chakarian JC, Ricard JD, Wittebole X, Chevalier S, Herbland A, Fartoukh M, Constantin JM, Tonnelier JM, Pierrot M, Mathonnet A, Beduneau G, Deletage-Metreau C, Richard JC, Brochard L, Robert R; FLORALI Study Group; REVA Network. High-flow oxygen through nasal cannula in acute hypoxemic respiratory failure. N Engl J Med. 2015 Jun 4;372(23):2185-96. doi: 10.1056/NEJMoa1503326. Epub 2015 May 17. PMID 25981908
- [Background] Grieco DL, Maggiore SM, Roca O, Spinelli E, Patel BK, Thille AW, Barbas CSV, de Acilu MG, Cutuli SL, Bongiovanni F, Amato M, Frat JP, Mauri T, Kress JP, Mancebo J, Antonelli M. Non-invasive ventilatory support and high-flow nasal oxygen as first-line treatment of acute hypoxemic respiratory failure and ARDS. Intensive Care Med. 2021 Aug;47(8):851-866. doi: 10.1007/s00134-021-06459-2. Epub 2021 Jul 7. PMID 34232336
- [Background] He Y, Zhuang X, Liu H, Ma W. Comparison of the efficacy and comfort of high-flow nasal cannula with different initial flow settings in patients with acute hypoxemic respiratory failure: a systematic review and network meta-analysis. J Intensive Care. 2023 May 10;11(1):18. doi: 10.1186/s40560-023-00667-2. PMID 37165464
- [Background] Ospina-Tascon GA, Calderon-Tapia LE, Garcia AF, Zarama V, Gomez-Alvarez F, Alvarez-Saa T, Pardo-Otalvaro S, Bautista-Rincon DF, Vargas MP, Aldana-Diaz JL, Marulanda A, Gutierrez A, Varon J, Gomez M, Ochoa ME, Escobar E, Umana M, Diez J, Tobon GJ, Albornoz LL, Celemin Florez CA, Ruiz GO, Caceres EL, Reyes LF, Damiani LP, Cavalcanti AB; HiFLo-Covid Investigators. Effect of High-Flow Oxygen Therapy vs Conventional Oxygen Therapy on Invasive Mechanical Ventilation and Clinical Recovery in Patients With Severe COVID-19: A Randomized Clinical Trial. JAMA. 2021 Dec 7;326(21):2161-2171. doi: 10.1001/jama.2021.20714. PMID 34874419
- [Background] Perkins GD, Ji C, Connolly BA, Couper K, Lall R, Baillie JK, Bradley JM, Dark P, Dave C, De Soyza A, Dennis AV, Devrell A, Fairbairn S, Ghani H, Gorman EA, Green CA, Hart N, Hee SW, Kimbley Z, Madathil S, McGowan N, Messer B, Naisbitt J, Norman C, Parekh D, Parkin EM, Patel J, Regan SE, Ross C, Rostron AJ, Saim M, Simonds AK, Skilton E, Stallard N, Steiner M, Vancheeswaran R, Yeung J, McAuley DF; RECOVERY-RS Collaborators. Effect of Noninvasive Respiratory Strategies on Intubation or Mortality Among Patients With Acute Hypoxemic Respiratory Failure and COVID-19: The RECOVERY-RS Randomized Clinical Trial. JAMA. 2022 Feb 8;327(6):546-558. doi: 10.1001/jama.2022.0028. PMID 35072713
- [Derived] Yaroshetskiy AI, Krasnoshchekova AP, Tkachenko FD, Rubashchenko AV, Zubarev DD, Konanykhin VD, Savelenok MI, Nosenko MM, Merzhoeva ZM, Avdeev SN. Gas composition and pressure in the hypopharynx during high-flow oxygen therapy through a nasal cannula in healthy volunteers with different breathing patterns. BMC Anesthesiol. 2025 Aug 23;25(1):416. doi: 10.1186/s12871-025-03267-9. PMID 40849448